CLINICAL TRIAL: NCT06334978
Title: The Effectiveness of Osteopathic Treatment in Cervical Whiplash.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Juan de Dios del Aljarafe de Sevilla (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1-2024
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Whiplash Injury of Cervical Spine; Osteopathia; Quality of Life; Chronic Pain Syndrome
Keywords: Whiplash Injury of Cervical Spine; Osteopathia; Quality of Life; Chronic pain; Functionality
MeSH Terms: conditions — Bone Diseases; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study was blinded: patients were unaware of the group to which they had been assigned. Patient evaluations at the start and end were performed by a physiotherapist different to the one performing the intervention, who was also unaware of the patient assignment. The same person performed all therapies for both the control and intervention groups and was unaware of the pre-intervention measurements. The statistician who analysed the data was also unaware of the group to which each patient belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Techniques used: the dog technique in flexion, scalene muscle energy technique, Jones' first rib adjustment, first rib trust in posterior subluxation, occipitomastoid thrust, Sutherland's posterior needle-scratch, SBS decompression, semi-direct thrust for the sacrum, Sutherland's sacrum, posterior occipital condyle thrust, SBS equilibration.
  Interventions: Other: Osteopathic intervention
- Control Group (No Intervention): Conventional treatment

INTERVENTIONS:
Other: Osteopathic intervention — The experimental group received the same treatment as the control group and one osteopathic intervention per week for the 21 days of the study (days 2, 9 and 16). Each session was performed on a different day from the conventional treatment to prevent interactions. The physiotherapist performed an osteopathic assessment involving a static/dynamic inspection and palpation and other osteopathic tests: Mitchell test, Quick Scanning, standing flexion (Piedallu) test, Gillet test, sphenobasilar synchondrosis (SBS) test, sutural palpation test and diaphragm test. Techniques used: the dog technique in flexion, scalene muscle energy technique, Jones' first rib adjustment, first rib trust in posterior subluxation, occipitomastoid thrust, Sutherland's posterior needle-scratch, SBS decompression, semi-direct thrust for the sacrum, Sutherland's sacrum, posterior occipital condyle thrust, SBS equilibration.
  Arms: Intervention Group

SUMMARY:
Introduction. Whiplash is common after road traffic accidents and affects millions of people worldwide; 50% develop chronic symptoms and 15% have their ability to work compromised. The aim of this study was to evaluate an osteopathic intervention in whiplash and determine whether pain, mobility and quality of life improve with respect to conventional treatment.

Methodology. A randomised, controlled clinical trial between 13/01/2021_10/08/2022 conducted at Hospital San Juan de Dios del Aljarafe. The control group followed the hospital's protocol, and the experimental group also received an osteopathic intervention. Statistical analysis: Statistical Package for the Social Sciences (SPSS-vs27.0); intra-subject comparison: Student's t-test for dependent samples, Wilcoxon's test; inter-group comparisons: Student's t-test for independent samples, Mann-Whitney U, chi-squared.

DETAILED DESCRIPTION:
A controlled randomised clinical trial (RCT) was carried out between 13 January 2021 and 10 August 2022 at the Hospital San Juan de Dios del Aljarafe, in Bormujos (Seville, Spain), a regional hospital covering a population of 300,000.

The main objective of the study was to determine whether the intervention proposed resulted in an improvement, in terms of pain, mobility and quality of life, compared with the local conventional treatment. The secondary objectives were to determine the decrease in medication and number of pain sites, as well as the influence of age and sex on the findings.

Patients were randomised to the control and intervention groups using the "Quickcalcs" program. The study was blinded: patients were unaware of the group to which they had been assigned. Patient evaluations at the start and end were performed by a physiotherapist different to the one performing the intervention, who was also unaware of the patient assignment. The same person performed all therapies for both the control and intervention groups and was unaware of the pre-intervention measurements. The statistician who analysed the data was also unaware of the group to which each patient belonged.

The inclusion criteria were: patients diagnosed with WAD grade II (Quebec classification), aged between 18 and 55 years, who started physiotherapy treatment less than 10 days prior to joining the trial, and who agreed to join the trial and provided informed consent. Patients with a history of neck pain in the previous three months (other than the whiplash), or with a prior history of WAD, or who had previously received osteopathic treatment for WAD, were excluded. Pregnant women, patients suspected to be simulating or exaggerating their symptoms for financial reasons, and those who presented difficulties carrying out the evaluation correctly due to their culture or a language barrier, were also excluded. Patients with a history of chest, head or upper limb surgery, those diagnosed with a neurological condition (such as congenital or diabetic polyneuritis, or any neurological condition), rheumatic alterations (such as osteoarthritis, arthritis, ankylosing spondylitis, etc.), malformations or surgical interventions that prevented correct conduct of the evaluation test and/or contraindications for the application of osteopathic and/or conventional treatment, were also excluded.

The sample size was calculated using the GRANMO calculator required for the main dependent variables, namely pain (visual analogue scale (VAS)) and quality of life (Whiplash Disability Questionnaire (WDQ)18 and Neck Disability Index (NDI))19. The highest of the three sample sizes calculated (that for WAD) was used, with 46 subjects being required in each group to detect a difference of 20 units or more, accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided comparison and assuming a common standard deviation of 25, a correlation coefficient between the initial and final measurement of 0.16 and a loss to follow-up of 10%.

A file was created for each patient containing their age, sex, height, weight, race and pharmacological treatment.

The initial (PRE) evaluation was carried out immediately prior to starting treatment (day 1) and the final (POST) evaluation, involving pressure algometry, inclinometry, VAS, NDI and WDQ, was carried out after treatment for 21 days. The WDQ was applied again at 4 weeks after completing treatment by way of a phone call.

The android application "Clinometer" was used to perform inclinometry20,21. The parameters flexion/extension and right and left cervical lateral flexion were measured with the patient sitting, with their feet on the floor and knees and hips at 90º, and a band was used to maintain the thoracic spine and arms attached to the rest while measurements were taken. Right and left cervical rotation were measured in a supine position.

An FPX 25 algometer (Wagner Instruments, Greenwich, CT, USA) was used to perform algometry22,23 bilaterally at two points: the mid-region of the anterior edge of the upper trapezius when sitting and the sternocleidomastoid when supine. The tip of the middle or index finger was placed under the trigger point and the tip of the algometer on the trigger point perpendicular to it. The pressure was increased gradually, at a rate of 1 kg/cm2/s, until the patient reported a change from a sensation of pressure to one of pain. Three measurements were performed at each point, with a rest time of 30 seconds between each measurement, and an additional 30 seconds before moving to the other point. The mean of the three measurements performed at each point was calculated. The algometer screen was placed facing the floor so that the results could not be seen until the measurement was complete.

The initial and final (PRE and POST) evaluations were recorded in a Google Form linked to each patient by way of their medical record number.

In addition, the patient completed a daily pain log using the VAS, indicated the location of the pain using a picture of the human body from an anteroposterior viewpoint, and recorded any medication taken, if required. This information was recorded twice daily, in the morning and evening, for 21 days.

The physiotherapist recorded the treatment administered in a document and, in the case of the experimental group, added the osteopathic tests and techniques used.

The standard treatment protocol for the Rehabilitation Service at the Hospital San Juan de Dios del Aljarafe is as follows: 30-minute sessions from Monday to Friday. Infrared radiation is applied to the cervical region for 15 minutes and session is completed by alternating massage and electrical currents (TENS) to the trapezii for 15 minutes. The patient is given a list of flexibility exercises for the cervical spine on the first day and performs them during the daily infrared treatment. This is the treatment for the control group.

The experimental group received the same treatment as the control group along with one osteopathic intervention per week for the 21 days of the study (days 2, 9 and 16). Each session was performed independently and on a different day from the manual therapy performed as part of the conventional treatment to prevent possible interactions, interferences and biases.

In order to adjust the treatment to the needs of each patient, based on their pathophysiology and the findings of the tests used, a personalised osteopathic intervention was proposed as part of the characteristics of a pragmatic study. Before selecting the techniques, the physiotherapist performed an osteopathic assessment involving a static/dynamic inspection and palpation and other osteopathic tests. The most common such tests were the Mitchell test, Quick Scanning, standing flexion (Piedallu) test, Gillet test, sphenobasilar synchondrosis (SBS) test, sutural palpation test and diaphragm test.

The techniques used most often were the dog technique in flexion, scalene muscle energy technique, Jones' first rib adjustment, first rib trust in posterior subluxation, occipitomastoid thrust, Sutherland's posterior needle-scratch, SBS decompression, semi-direct thrust for the sacrum, Sutherland's sacrum, posterior occipital condyle thrust, SBS equilibration.

The statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) version 27.0. For the comparative intra-subject analysis, Student's t-test was used for dependent variables (those with a normal distribution) and Wilcoxon's test for those with a non-normal distribution. Similarly, Student's t-test for independent samples and the Mann-Whitney U test were used to compare the results for the various dependent variables, depending on whether the distribution thereof was normal or not. The chi-squared test (sex as qualitative variable), Student's t-test for independent samples (variables with a normal distribution) and the Mann-Whitney U test (non-normal distribution) were used to evaluate the characteristics of the samples from each group. Statistical significance: p<0.05.

The ethical principles for medical research involving human subjects set out in the Declaration of Helsinki, and its updates, and Law 14/2007, of 03 July, on biomedical research, were taken into consideration This trial was approved by the Research Ethics Committee of the Virgen del Rocío University Hospital (internal code: 2015-N-18). All participants received information prior to the study and provided written informed consent. The treatment, communication and transfer of participants' personal data is in accordance with Organic Law 3/2018, of 05 December, on personal data protection and the guarantee of digital rights.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with WAD grade II (Quebec classification),
* aged between 18 and 55 years,
* who started physiotherapy treatment less than 10 days prior to joining the trial,
* and who agreed to join the trial and provided informed consent.

Exclusion Criteria:

* Patients with a history of neck pain in the previous three months (other than the whiplash),
* or with a prior history of WAD,
* or who had previously received osteopathic treatment for WAD,
* Pregnant women,
* patients suspected to be simulating or exaggerating their symptoms for financial reasons,
* those who presented difficulties carrying out the evaluation correctly due to their culture or a language barrier.
* Patients with a history of chest, head or upper limb surgery,
* those diagnosed with a neurological condition (such as congenital or diabetic polyneuritis, or any neurological condition),
* or rheumatic alterations (such as osteoarthritis, arthritis, ankylosing spondylitis, etc.),
* or malformations or surgical interventions that prevented correct conduct of the evaluation test
* and/or contraindications for the application of osteopathic and/or conventional treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Cervical Pain | 3 measurements: Just before starting the study, at 21 days and at 4 weeks.
  Pain measured with the "visual analogue scale" (scale: 0-10)
Quality of life in Whiplash Disability | 3 measurements: Just before starting the study, at 21 days and at 4 weeks.
  Quality of life measured with the Whiplash Disability Questionnaire (scale: 0-130)
Functionality-Neck Disability Index | 3 measurements: Just before starting the study, at 21 days and at 4 weeks.
  Functionality measured with the Neck Disability Index (scale: 0-100). Each question is measured on a scale from 0 (no disability) to 5 (most disabled), and an overall score of 100 is calculated by adding the score for each item and multiplying by two. A higher NDI score means greater perceived patient disability due to neck pain. The "minimally clinically important change" by patients has been found to be 5 or 10%.

SECONDARY OUTCOMES:
Number of sites | 4 measurements: Just before starting the study, at 7 days, at 21 days and at 4 weeks.
  Number of sites whit pain
Number of analgesics | 4 measurements: Just before starting the study, at 7 days, at 21 days and at 4 weeks.
  Number of analgesics

OTHER OUTCOMES:
Measuring mobility using inclinometry | 2 measurements: Just before starting the study, at 4 weeks
  For inclinometry, the Android App: Clinometer was used. The parameters of flexion (scale 0º-45º), extension (scale 0º-45º), lateral inclination (scale 0º-45º) and rotation (scale 0º-80º). 0º being no mobility and 45º or 80º being the best mobility.
Measurement of pressure pain using algometry | 2 measurements: Just before starting the study, at 4 weeks
  For algometry, the model FPX 25 algometer (Wagner Instruments, Greenwich, CT, USA) was used. Scale 0-100; unit:Ibf. The greater the pressure exerted, the better the person tolerates the pain, so the result is more positive. It was measured at two points bilaterally: the middle region of the anterior edge of the upper trapezius in sitting position and the sternocleidomastoid.

CONTACTS AND LOCATIONS:
Overall Officials: José Larios Ortega, Graduate, Principal Investigator — Physiotherapy Unit. Rehabilitation Service. Hospital San Juan de Dios del Aljarafe.
Locations (1):
- María Victoria RUIZ ROMERO, Bollullos de la Mitación, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No
We will not be shared with other researchers individual participant data.